CLINICAL TRIAL: NCT02697487
Title: UTSW Depression Cohort: A Longitudinal Study of Depression
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU 092015-049
Record Dates: First submitted 2016-02-23; First posted 2016-03-03 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Depression; Other Diagnoses, Comorbidities, and Complications
Keywords: Depression; Cohort
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biospecimens being studied is as follows:
  1. Blood
  2. Normal Tissue
  3. Saliva
  4. Urine
  5. Stool
  6. Clinical waste products to include surgical waste tissue samples, placenta samples, and biopsy samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- No Treatment: This is a longitudinal observational study involving individuals who are depressed, depressed with other comorbidities and non-depressed individuals. The primary aim of this study is to describe the longitudinal course of illness and real world treatment outcomes for depressed patients receiving routine care from their providers. Health outcomes and biospecimens along with the functional and economic burden of depression will be characterized and compared amongst three groups: (1) depressed patients, (2) depressed patients with comorbid illnesses, and (3) non-depressed patients.
  Interventions: Other: No treatment

INTERVENTIONS:
Other: No treatment — This is an observational study with no intervention.

SUMMARY:
This is a longitudinal observational study (via electronic records and biospecimens) designed to utilize health IT advances to collect information from patients undergoing routine care. This information will be stored in a database. Patients undergoing routine care from their providers will be invited to participate in the UTSW Depression Cohort. After obtaining informed consent, the CDRCC team will collect information from available sources and store it in a secure UT Southwestern network database protected by a security firewall. A schematic representation of this information processing is shown in the figure contained in section 3 of the protocol. As part of the UTSW Depression Cohort, patients will allow banking of their specimens. Specimens which are banked may include blood or blood products, urine, tissue samples, saliva, stool samples or clinical waste products. The study will only enroll participants comfortable with providing specimens. As the goal of the UTSW Depression Cohort is to create a national database, CDRCC will engage with patients, providers, and researchers at local, regional, and national levels. A large number of medical providers are already screening patients for depression. Structured instruments like PHQ-2 or PHQ-9 are often used. Hence, the CDRCC will seek collaborations with local, regional and national partners so that information contained in their health IT initiatives can be included in the this database. Due to the clinical nature of information collected, the investigators anticipate marked heterogeneity in the variables and amount of data collected. Database architects will utilize big data (large volumes of information from diverse sources with variable degrees of quality and complexity) tools to structure the registry so that additional variables can be added, as needed. The CDRCC team will maintain a detailed codebook of variables collected in the database. All statistical analyses will be conducted only on de-identified data. Researchers may obtain access to this de-identified data by following procedures established by the CDRCC, which include obtaining IRB approval.

DETAILED DESCRIPTION:
This is a longitudinal observational study designed to utilize health IT advances to collect information from patients undergoing routine care. This information will be collected as part of routine care and stored in a database for research purposes. Patients undergoing routine care from their providers will be invited to participate in the UTSW Depression Cohort. After obtaining informed consent, the CDRCC team will collect information from sources outlined in background section of protocol and store it in a secure UT Southwestern network database protected by a security firewall. A schematic representation of this information processing is shown on page 7 of the protocol. The CDRCC team will also collect specimens which are obtained as part of standard of care and are beyond the amount needed for routine clinical care. For research-only purposes, CDRCC team will also collect blood, saliva, stool and urine specimens at regular intervals described in subsequent section with the consent of study participant.

Clinics or health care facilities collaborating with CDRCC will approach their patients to participate in this cohort. Research staff from UTSW or staff at these clinics (or health care facilities) who have received training on how to obtain informed consent will then ask interested patients to sign the IRB-approved Informed Consent and HIPAA authorization documents. Initially, the Informed Consent and HIPAA authorization will be documented on paper, and these documents will be scanned and stored in the master log of the Cohort database in addition to securely storing the paper copy. In the future, patients will be asked to complete Informed Consent and HIPAA authorization documents using computers or handheld electronic devices (including signatures). Paper documents will be made available to those who prefer and request them. Staff from CDRCC will be available either in person, by email, or by phone to answer any questions that arise during the informed consent process that cannot be answered by clinic staff. If patients are under the age of 18, they will provide assent, and a parent or LAR will provide consent. The CDRCC will also develop materials in print and electronic format to publicize the UTSW Depression Cohort. Other patients or healthy individuals who are not involved with a CDRCC collaborator can also join the registry if they complete the informed consent process. The UTSW Depression Cohort will include comprehensive information collected as part of routine care by the patient's provider(s). During routine care at their medical providers' offices, patients may fill out screening questionnaires and self-rated behavioral health assessments, provide medical and psychiatric history, undergo laboratory tests, electrocardiogram (EKG), radiologic or other clinically relevant investigations and be given treatment recommendations. Some of the self-rated assessments completed as part of measurement based care may include Patient Health Questionnaire 2 (PHQ-2), Patient Health Questionnaire 9 (PHQ-9), Patient Adherence Questionnaire (PAQ), Frequency, Intensity, and Burden of Side Effects Rating (FIBSER), Generalized Anxiety Disorder 7 (GAD-7), Concise Associated Symptoms Tracking - Self-Report Scale (CAST-SR), Pain Frequency, Intensity, and Burden Scale (P-FIBS), Concise Health Risk Tracking Scale (CHRT), and Alcohol and Drug usage screen. The information in the Cohort database will be stored indefinitely unless a participant requests the principal investigator to remove his/her name and associated information.

Research only assessments As part of the UTSW Depression Cohort, participants will undergo diagnostic assessment using MINI International Neuropsychiatric Interview, Version 7.0 for DSM-5 (MINI) and complete self-report research assessments for psychiatric symptoms and psychosocial functioning. These research only assessments will add 60-90 minutes to the visit duration.

Specimen banking:

As part of the UTSW Depression Cohort, patients will allow banking of their specimens. The study will only enroll participants comfortable with providing specimens. Of course, like with any other study procedure, those not comfortable with providing specimens will not be enrolled in this study. Specimens which are banked may include blood or blood products, urine, stool samples, tissue samples, saliva or clinical waste products. Clinical waste products include surgical waste tissue samples, placenta samples and biopsy samples. Once a sample is collected, all identifying information will be removed, and it will be given a unique code. The information linking this unique code to a patient's identifying information will be stored in the master log. Samples will be stored appropriately in the CDRCC freezers located in the north campus building of UT Southwestern. Samples will be overseen by CDRCC research personnel. A sample will be stored indefinitely until the sample runs out or it is destroyed.

Blood and blood products- Blood will be obtained by venipuncture performed by personnel with phlebotomy training.

Adult blood draws will not exceed the following:

Patient weight Maximum Volume per 24 hour Maximum Volume per Month Kilograms Pounds Milliliters Milliliters 51-60 112-132 112-120 224-240 61-65 134-143 122-130 244-260 68-70 145-154 132-140 264-280 71-75 156-185 142-150 284-300 76-80 167-176 152-160 304-360 81-85 178-187 162-170 324-340 86-90 189-198 172-180 344-360 91-95 200-209 182-190 364-380 96-100 211-220 192-200 384-400

Pediatric blood draws will not exceed:

Patient weight Maximum Volume per 24 hour Maximum Volume per Month Kilograms Pounds Milliliters Milliliters <0.9 <2 3 12 0.9-1.8 2-4 4.5 18 1.9-2.7 4-6 6 24 2.8-3.6 6-8 7.5 30 3.7-4.5 8-10 10.5 42 4.6-6.8 10-15 15 60 6.9-9.1 16-20 30 120 9.2-11.4 21-25 30 120 11.5-13.6 26-30 30 120 13.7-15.9 31-35 30 120 16.0-18.2 36-40 30 120 18.3-20.5 41-45 60 240 20.6-22.7 46-50 60 240 22.8-25.0 51-55 60 240 25.1-27.3 56-60 60 240 27.4-29.5 61-65 75 300 29.6-31.8 66-70 90 360 31.9-34.1 71-75 90 360 34.2-36.4 76-80 90 360 36.5-38.6 81-85 90 360 38.7-40.9 86-90 90 360 41.0-43.2 91-95 90 360 43.3-45.5 96-100 90 360

Blood may be obtained as a single blood draw, which may be a patient's only collection. Patients may be contacted to provide similar specimens at intervals around every 3-4 months for over 5-10 years (for a total of 40 blood draws). Collections will be restricted by the maximum safe volumes outlined above for both adult and pediatric participants. If being obtained in a clinical setting, clinical care specimens will take precedence over research specimens. If specimens are obtained during the course of clinical care, a safe volume will be determined in conjunction with treating physicians, but will not exceed the above table.

Saliva- Saliva will be collected into the Oragene DNA and/or RNA self-collection kit and stored at room temperature until DNA isolation.

Urine- Urine samples will be collected in sterile urinalysis cups and 10 mL aliquots will be frozen at -80°C in conical tubes.

Stool- Stool samples will be collected once or possibly over time in conjunction with blood draws described above in sterile 50 ml conical tubes and will be frozen at -80°C.

Clinical waste products- Samples obtained could include: a. surgical waste tissue samples; b. placenta samples; and c. biopsy samples. These samples will be obtained as a part of standard of care. Procedures involving these sample collections will be done by trained physicians and medical technicians only. The tissue that will be used for research is the tissue that would normally be discarded. After providing informed consent, study participants may allow study personnel to collect these clinical waste products from the clinical sites. The clinical waste product will then be transported to CDRCC on ice for storage. These samples will be de-identified, stored and used for future research. There will be no cost or compensation to the patients for donating this tissue to CDRCC.

The intended use of these samples is to enable future research into the diagnostics, prognostics and biologic understanding of depression. The samples will be primarily used by investigators affiliated with UT Southwestern, but will also be released to public and private collaborators in a HIPAA compliant fashion (i.e., de-identified). Development of cell lines and DNA libraries may occur with these samples. Samples may be used by investigators not affiliated with UT Southwestern if they are collaborating with a UTSW investigator. Also, samples may be used by colleagues at other institutions who are conducting their own IRB -approved research. Furthermore, de-identified samples can be provided to collaborators in industry if appropriate technology transfer agreements are in place. Samples sent to investigators or private entities outside of UT Southwestern will have a charge associated with them based on sample cost and projected use of the samples. Any specimen or data can be released to collaborators (outlined above) as long as it is released in a HIPAA compliant fashion (i.e., de-identified).

The investigators will obtain an IRB approval letter and maintain a current record of the Federal Wide Assurance (FWA) for an IRB at another medical center if data and specimens are sent from human cell banks at UT Southwestern to another medical center. If an investigator at another medical center receives data and specimens from our Cohort at UT Southwestern, the investigator will maintain documentation that (a) the recipient of samples from CDRCC acknowledges that the conditions for use of the research material are governed by the IRB at UT Southwestern in accordance with 45 CFR 46, (b) the recipient agrees to comply fully with all such conditions and to report promptly to the CDRCC at UT Southwestern any proposed changes in the research project, (c) the recipient remains subject to applicable State or local laws or regulations and institutional policies which provide additional protections for human subjects, and (d) the research material may be utilized only in accordance with the conditions stipulated by the IRB at UT Southwestern. Any additional use of this material requires prior review and approval by the IRB at UT Southwestern and, where appropriate, by an IRB at the recipient site, which must be convened under an applicable OHRP-approved Assurance. Non-UT Southwestern recipients of samples will be charged a usual and customary fee for the sample to cover procurement costs.

Under the supervision of the principal investigator of CDRCC, two different subcommittees will oversee the different aspects of the UTSW Depression Cohort: data management committee and executive committee. The data management committee will be tasked with managing the flow of information into and out of the Cohort database, maintaining the codebook of variables, developing big data tools (as mentioned in specific aim 3), and ensuring consistency of data collection and quality. The executive committee will be tasked with all other responsibilities related to the registry like establishing collaborations with providers, reviewing research proposals, and providing access to the cohort data for qualified researchers.

All procedures will be conducted as part of a patient's routine medical care except for collection of research-only blood, urine, and saliva specimens as described above. This study does not involve any interventions.

ELIGIBILITY:
Inclusion Criteria:

* Participants ages 10 - 89 years who speak English or Spanish (consent and HIPAA authorization forms will be translated in Spanish for mono-lingual Spanish-speaking only participants).
* Provide informed consent (parent or LAR for participants aged 10 to 17).

Exclusion Criteria:

* Participants who do not speak English or Spanish.
* Participants who are less than 10 or greater than 89 years old.

Ages: 10 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The following groups are being targeted for this observational study:
  1. depressed patients,
  2. depressed patients with comorbid illnesses, and
  3. non-depressed patients.
Sampling Method: Non-Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2016-02; Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

PRIMARY OUTCOMES:
Changes in depression severity as measured by 9-item Patient Health Questionnaire | Change from Baseline to 10 years
  Changes in depression severity will be measured by 9-item Patient Health Questionnaire. PHQ-9 score ranges from 0-27, higher score indicates sever depression.
  Minimal depression 0-4 Mild depression 5-9 Moderate depression 10-14 Moderately severe depression 15-19 Severe depression 20-27

SECONDARY OUTCOMES:
Changes in functioning as measured by 5-item Work Social Adjustment Scale in participants with and without depression. | Change from Baseline to 10 years
  Changes in functioning will be measured by 5-item Work Social Adjustment Scale (WSAS).5-item Work Social Adjustment Scale ranges from 0 to 40.
  WSAS Score >20 appears to suggest moderately severe or worse psychopathology Scores between 10 and 20 are associated with significant functional impairments but less severe clinical symptomatology.
  Scores <10 appear to be associated with subclinical population

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes